CLINICAL TRIAL: NCT00233532
Title: A Prospective, Open-Label Study to Evaluate the Effect of an Escalating Dose Regimen of Trandolapril on Blood Pressure in Treatment-Naïve and Concurrently Treated Hypertensive Patients (TRAIL)
Brief Title: Canadian Study of Trandolapril on Blood Pressure in Hypertensive Patients (TRAIL)
Acronym: TRAIL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Anita Vanjaka, Clinical Research Manager, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CANA-03-003
Record Dates: First submitted 2005-09-13; First posted 2005-10-06 (Estimated); Last update posted 2008-07-22 (Estimated); Status verified 2008-07

CONDITIONS: Hypertension
Keywords: Hypertension; Trandolapril
MeSH Terms: conditions — Hypertension | interventions — trandolapril; Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other)
  Interventions: Drug: Trandolapril
- 2 (Other)
  Interventions: Drug: Trandolapril
- 3 (Other)
  Interventions: Drug: Trandolapril

INTERVENTIONS:
Drug: Trandolapril — 0.5, 1,2,4mg/once daily/ for 26 weeks (If BP was not controlled, dose was escalated to the next higher dosage every 4-5 weeks).
  Other Names: ABT-TARKA; trandolapril/verapamil; TARKA

SUMMARY:
The TRAIL study was conducted to examine the effects of escalating doses of an ACE inhibitor, trandolapril, on lowering blood pressure in Stage 1-2 hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1 or 2 Hypertension

Exclusion Criteria:

* Uncontrolled diabetes
* Subject has a hypersensitivity to ACE inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2004-03; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Effectiveness of escalating dose regimen of trandolapril in controlling blood pressure | 14 weeks

SECONDARY OUTCOMES:
Changes in blood pressure, safety. | 14 and 26 weeks
BP mmHg incremental and absolute change | 14 and 26 weeks
Adverse events | Throughout 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information 1-800-633-9110, Study Director — Abbott